CLINICAL TRIAL: NCT03899324
Title: A Randomized Double-blind Placebo-controlled Multicenter Proof-of-concept Trial to Assess the Efficacy and Safety of Bumetanide in Parkinson's Disease
Brief Title: Evaluation of the Efficacy and Safety of Bumetanide in Parkinson's Disease
Acronym: CUREPARK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: B&A Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUREPARK/OP105018.BAT
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Experimental Bumetanide (Experimental): bumetanide with a titration period
  Interventions: Drug: Bumetanide white, oblong, scored tablet
- Group 2: Placebo comparator (Placebo Comparator): placebo intake identically to group 1
  Interventions: Drug: Placebo white, oblong, scored tablet

INTERVENTIONS:
Drug: Bumetanide white, oblong, scored tablet — Bumetanide with a titration period
  Arms: Group 1: Experimental Bumetanide
Drug: Placebo white, oblong, scored tablet — placebo intake identically to group 1
  Arms: Group 2: Placebo comparator

SUMMARY:
This is multicentre, proof of concept, randomized, double-blind, parallel-group, placebo-control study in 40 Parkinson's Disease (PD) patients. Patients will be randomized in 2 groups receiving Bumetanide or placebo for 4 months:

* Group 1 (20 PD patients): bumetanide
* Group 2 (20 PD patients): placebo intake identically to group 1.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease fulfilling the UK Parkinson's Disease Brain Bank (UKPDSBB) criteria (cf. Appendix VII)
2. 40 < Age < 80 years old
3. Hoehn & Yahr 1.5-4 (OFF stage)
4. Walking and balance or freezing ≥ 1in the MDS-UPDRS II
5. Motor fluctuation defined by a score ≥ 1 on the item "time spent in the OFF state" of the MDS-UPDRS IV
6. Dose of L-DOPA ≥ 150 mg/d (concomitant treatment)
7. PD medications regimen stable for at least 3 months
8. Patients expected to remain on stable doses of PD medications during all the study
9. Covered by Health Insurance System
10. Able to understand and to sign the informed consent prior to selection
11. Negative pregnancy test at screening
12. Blood Pressure (BP) and Heart Rate (HR) considered Non Clinicaly Significant (NCS) by investigators
13. Electrocardiogram (ECG) recording on a 12-lead ECG considered NCS by investigators
14. Laboratory parameters within the normal range of the laboratory. Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator

Exclusion Criteria:

1. Atypical parkinsonism or drug-induced parkinsonism
2. Cognitive impairment (MMSE ≤ 24)
3. Active psychiatric disorder (mood disorders, hallucinations or delirium with strong functional impact and not controlled by medication or which happened during the last 3 months before inclusion)
4. Treatment by Deep Brain Stimulation or continuous infusion of apomorphin/dopa gel
5. Renal or hepatic insufficiency
6. Electrolyte disturbances
7. A corrected QT (QTcF) interval >450ms for male or >470ms for female on the electrocardiogram
8. Any medical condition that might interfere with the protocol except those defined in Section 5.3
9. Contraindications to bumetanide : persistent anuria, hepatic encephalopathy included coma
10. Women pregnant, nursing or of childbearing age without effective contraception. Patients should not be enrolled if they plan to become pregnant during the time of study participation
11. Patient unable to attend scheduled visits or to comply to the protocol
12. Patient under legal guardianship or judicial protection
13. Patient in the exclusion period of another protocol
14. No possibility of contact in case of emergency
15. Known allergic reactions induced by Burinex (Bumetanide)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the change from baseline (V2) to endpoint (V5) in the MDS-UPDRS III motor score, evaluated 1 hour after the intake of the study treatment (Bumetanide or placebo) in patients in the OFF state. | Between Day 1 and Day 120

SECONDARY OUTCOMES:
Change from V2 to V5 of the MDS-UPDRS part III and part I measured in a patient in the ON state. | Between Day 1 and Day 120
  Movement Disorder Society Unified Parkinson's Disease Rating Scale
Change of scores of the MDS-UPDRS part II, III and IV during the trial, at D1 (V2), D30 (V3), D60 (V4) and D120 (V5). | Day 1, Day 30, Day 60, Day 120
  Movement Disorder Society Unified Parkinson's Disease Rating Scale
Stand-Walk-Sit test at D1 (V2), D30 (V3), D60 (V4) and D120 (V5). | Day 1, Day 30, Day 60, Day 120
Number of adverse events collected at each visit and phone calls. | Throughout the completion of the study, from Day 1 to Day 135

OTHER OUTCOMES:
Unified dyskinesia rating scale at D1 (V2), D30 (V3), D60 (V4) and D120 (V5). | Day 1, Day 30, Day 60, Day 120
Awaken time spent in the OFF state, in the ON state with and without dyskinesia. | Between Day 0 (Screening) and Day 1 (V2), then between Day 60 (V4) and Day 120 (V5)
Patient's Clinical Global Impression (CGI) score at D1 (V2), D30 (V3), D60 (V4) and D120 (V5). | Day 1, Day 30, Day 60, Day 120

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nantes, Nantes, France

REFERENCES:
- [Background] Damier P, Hammond C, Ben-Ari Y. Bumetanide to Treat Parkinson Disease: A Report of 4 Cases. Clin Neuropharmacol. 2016 Jan-Feb;39(1):57-9. doi: 10.1097/WNF.0000000000000114. PMID 26757306
- [Background] Lozovaya N, Eftekhari S, Cloarec R, Gouty-Colomer LA, Dufour A, Riffault B, Billon-Grand M, Pons-Bennaceur A, Oumar N, Burnashev N, Ben-Ari Y, Hammond C. GABAergic inhibition in dual-transmission cholinergic and GABAergic striatal interneurons is abolished in Parkinson disease. Nat Commun. 2018 Apr 12;9(1):1422. doi: 10.1038/s41467-018-03802-y. PMID 29651049